CLINICAL TRIAL: NCT06874179
Title: Effects of Oropharyngeal-topical and Intravenous Lidocaine on the Optic Nerve Sheath Diameter Changes After Endotracheal Intubation: a Randomized Controlled Clinical Study
Brief Title: Oropharyngeal Vs Intravenous Lidocaine Effects on Optic Nerve Sheath Diameter After Intubation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, Ass.Prof.Dr. İsmail Aytaç, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: TABED 1-24-831
Record Dates: First submitted 2025-01-14; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-01

CONDITIONS: Endotracheal Intubation During Surgery; Optic Nerve Sheath Diameter
Keywords: endotracheal intubation; optic nerve sheath diameter; lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded (Participants and Outcome Assessors)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Pre-intubation oropharyngeal topical %10 lidocaine (Experimental): Participants will receive 10% lidocaine spray topically to the oropharynx before intubation.
  Interventions: Diagnostic Test: Optic nerve sheath diameter measurement 0; Diagnostic Test: optic nerve sheath diameter measurement 1; Diagnostic Test: optic nerve sheath diameter measurement 2; Diagnostic Test: optic nerve sheath diameter measurement 3; Procedure: Pre-intubation oropharyngeal topical %10 lidocaine
- Group B: Pre-intubation intravenous %2 lidocaine (Experimental): Participants will receive 2% lidocaine intravenously before intubation.
  Interventions: Diagnostic Test: Optic nerve sheath diameter measurement 0; Diagnostic Test: optic nerve sheath diameter measurement 1; Diagnostic Test: optic nerve sheath diameter measurement 2; Diagnostic Test: optic nerve sheath diameter measurement 3; Procedure: Pre-intubation intravenous %2 lidocaine

INTERVENTIONS:
Diagnostic Test: Optic nerve sheath diameter measurement 0 — optic nerve sheath diameter (ONSD) measured via ultrasonography before intubation
Diagnostic Test: optic nerve sheath diameter measurement 1 — optic nerve sheath diameter measurement 1 via ultrasonography after intubation 1st minute
Diagnostic Test: optic nerve sheath diameter measurement 2 — optic nerve sheath diameter measurement via ultrasonography after intubation 5th minute
Diagnostic Test: optic nerve sheath diameter measurement 3 — optic nerve sheath diameter measurement via ultrasonography after intubation 10th minute
Procedure: Pre-intubation oropharyngeal topical %10 lidocaine — Pre-intubation oropharyngeal topical %10 lidocaine
  Arms: Group A: Pre-intubation oropharyngeal topical %10 lidocaine
Procedure: Pre-intubation intravenous %2 lidocaine — Pre-intubation intravenous %2 lidocaine
  Arms: Group B: Pre-intubation intravenous %2 lidocaine

SUMMARY:
This study aims to evaluate the effects of pre-intubation oropharyngeal topical lidocaine on optic nerve sheath diameter (ONSD) post-endotracheal intubation. The study will measure the ONSD using ultrasonography before intubation, and at 1, 5, and 10 minutes post-intubation. The results will be compared between patients receiving %10 lidocaine topically and %2 intravenous lidocaine.

DETAILED DESCRIPTION:
Increased intracranial pressure (ICP) is a critical condition that requires early and accurate assessment. Traditional invasive ICP monitoring techniques, such as lumbar puncture and intracranial pressure monitoring devices, carry significant risks. Optic nerve sheath diameter (ONSD) measurement via ultrasonography is a non-invasive method that reflects increased ICP.

Patients will be divided into two groups: Group A will receive %10 topical oropharyngeal lidocaine, and Group B will receive %2 intravenous lidocaine. The primary aim of the study is to evaluate the impact of lidocaine on ONSD at 1, 5, and 10 minutes post-intubation and to compare the effects on the two groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I or II
* Age 18-65 years
* BMI 18-30
* No history or expected difficult intubation
* No glaucoma or ocular pathology
* No intracranial pressure increase

Exclusion Criteria:

* ASA class III and above
* Obesity (BMI > 30)
* Difficult intubation history or risk
* Glaucoma or other ophthalmic pathology
* History of intracranial pressure increase or prior ophthalmic/intracranial surgery
* Preoperative sedation
* Active malignancy or ongoing radiotherapy/chemotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter 0 | Before intubation
  optic nerve sheath diameter (ONSD) measured via ultrasonography before intubation
Optic nerve sheath diameter 1 | 1 minute after intubation
  optic nerve sheath diameter (ONSD) measured via ultrasonography 1 minute after intubation
Optic nerve sheath diameter 2 | 5 minutes after intubation
  Optic nerve sheath diameter (ONSD) measured via ultrasonography 5 minutes after intubation
0ptic nerve sheath diameter 3 | 10th minutes after intubation
  0ptic nerve sheath diameter (ONSD) measured via ultrasonography 10th minutes after intubation

SECONDARY OUTCOMES:
Postoperative sore throat | 1 hour after recovery room admission
  Postoperative sore throat is evaluated with Visual Analog scale

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Aytaç, Ass. Prof, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data (IPD) will be made available upon request to scientific committees or researchers for further analysis, subject to ethical and privacy considerations.